CLINICAL TRIAL: NCT05310864
Title: Comparison of the Distance Between the Femoral Artery and Veins in Anatomic Position, Abduction-exorotation and Lower Limb Flexion Position (Frog Leg Position): Observational Study Using Ultrasonography in Malay Race Adult in Indonesia
Brief Title: Comparison of the Distance Between the Femoral Artery and Veins in Various Position in Malay Race Adult
Status: Completed | Type: Observational
Sponsor: Aldy Heriwardito (Other)
Responsible Party: Sponsor-Investigator, Aldy Heriwardito, Principal Investigator, Indonesia University
Organization: Indonesia University (Other)
Other Study IDs: IndonesiaUAnes395
Record Dates: First submitted 2022-03-14; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Femoral Artery and Vein Distance; Anatomic
Keywords: femoral artery; femoral vein; ultrasonography; Frog leg position; abduction-exorotation position

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to compare the distance between femoral artery and vein in frog position, abduction-exorotation position and anatomical position.

DETAILED DESCRIPTION:
The incidence of unintentional arterial puncture during cannulation of femoral vein was high(20-50%). The addition of knee flexion to abcudtion-exorotation position (frog position) have been shown to increase the cross sectional area of femoral vein. The purpose of this study is to compare the distance between femoral artery and vein in frog position, abduction-exorotation position and anatomical position.

This study is an analytical observational study with cross sectional design within one grup with repeated measurement. The distance between artery and vein was measured in three position. The measurement was taken twice for each position. First picture was taken by one operator and one ultrasonography for all patient. Then another operator measured the distances with caliper feature on the ultrasonograph.

ELIGIBILITY:
Inclusion Criteria:

1. Malay race adult 18-60 years old
2. Agree to participate in the study and undergoing femoral vein cannulation
3. Normal weight with IMT 19-25 kg/m2

Exclusion Criteria:

1. Previous cannulation on the same vein
2. Femoral vein catheter has been placed
3. Anatomical variation (artery-venous malformation, venous or artery branch at 2 cm inferior to inguinal ligament)
4. Abdominal distention
5. Femoral vein thrombosis
6. Hypotension (Mean Arterial Pressure <65 mmHg, or using vasopressor or inotrope)

Drop out Criteria:

1. Anatomical abnormalities of femoral vein or artery visualized using ultrasonography examination
2. Fail to visualize femoral vein or artery using ultrasonography for two minutes, operated by trained personnel and declared competent by cardiovascular anesthesiologist consultant
3. Patient not cooperative during procedure, hence, unable to maintain limb position for more than 2 minutes in any position examined
4. Patients with right femur fracture

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All Malay race adult seeking for medication in Ciptomangunkusumo Hospital who agree to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
The distance between femoral vein and artery in millimeter | one day at diagnosis day
  The distance between femoral vein and artery in frog leg position, abduction-exorotation position, and anatomical position

CONTACTS AND LOCATIONS:
Overall Officials: Aldy Heriwardito, Doctor, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia